CLINICAL TRIAL: NCT02041650
Title: Plaque Erosion: A New in Vivo Diagnosis and Paradigm Shift in the Treatment of Patients With Acute Coronary Syndrome
Brief Title: Paradigm Shift in the Treatment of Patients With ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yu Bo (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Yu Bo, Director of Cardiology of The 2nd Affiliated Hospital of Harbin Medical University, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0186; ISSBRIL0186 (Other: HarbinMU)
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with ACS treated medically (Other)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor

SUMMARY:
This protocol describes a pilot study intended to test the hypothesis that patients with acute coronary syndrome (ACS) caused by plaque erosion can be stabilized by effective antithrombotic treatment without stent implantation, thereby avoiding both early and late complications related to percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women >18 years of age and < 75 years of age
* Patients undergo cardiac catheterization for ACS. Patients with STEMI, NSTEMI, and UAP will be included. STEMI will be defined as continuous chest pain for >30 minutes, arrival at the hospital within 12 hours from chest pain onset, ST-segment elevation >0.1 mV in at least two contiguous leads, or new left bundle-branch block on the 12-lead electrocardiogram (ECG), and elevated cardiac markers (troponin T/I or creatine kinase-MB). NSTEMI will be defined as a progressive crescendo pattern of angina or angina at rest, in the absence of ST-segment elevation on the 12-lead ECG, with elevated cardiac markers. UAP will be defined as new onset angina, progressive crescendo pattern of angina, or angina at rest.
* Culprit lesion located in a native coronary artery
* TIMI flow grade 3 and diameter stenosis < 70% on angiogram
* Definite erosion defined by OCT
* Patients able to provide written informed consent

Exclusion Criteria:

Left ventricular ejection fraction < 30%.

* Life expectancy < 1 year.
* Contraindication to the contrast media.
* Creatinine level > 2.0 mg/dL or end-stage kidney disease.
* Serious liver dysfunction.
* Patients with hemodynamic or electrical instability (including shock).
* Any contraindication against the use of ticagrelor.
* Investigator considers the patient is not suitable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Reduction of thrombus burden by OCT | 30 days
  The efficacy will be assessed by 50% reduction in thrombus burden by OCT at 1 month.

SECONDARY OUTCOMES:
Cardiovascular adverse events | 30 days and 12 months
  In patients treated conservatively, the safety objectives are to evaluate the occurrence of any adverse events during1 month follow up (re-infarction, re-hospitalization, revascularization by PCI or CABG, cardiac death, stoke, and major bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD, PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

REFERENCES:
- [Derived] Seegers LM, Yeh DD, Wood MJ, Yonetsu T, Minami Y, Araki M, Nakajima A, Yuki H, Ako J, Soeda T, Kurihara O, Higuma T, Kimura S, Adriaenssens T, Nef HM, Lee H, McNulty I, Sugiyama T, Kakuta T, Jang IK. Cardiovascular Risk Factors and Culprit Plaque Characteristics in Women With Acute Coronary Syndromes. Am J Cardiol. 2023 Nov 15;207:13-20. doi: 10.1016/j.amjcard.2023.08.152. Epub 2023 Sep 16. PMID 37722196
- [Derived] Zeng M, Zhao C, Bao X, Liu M, He L, Xu Y, Meng W, Qin Y, Weng Z, Yi B, Zhang D, Wang S, Luo X, Lv Y, Chen X, Sun Q, Feng X, Gao Z, Sun Y, Demuyakor A, Li J, Hu S, Guagliumi G, Mintz GS, Jia H, Yu B. Clinical Characteristics and Prognosis of MINOCA Caused by Atherosclerotic and Nonatherosclerotic Mechanisms Assessed by OCT. JACC Cardiovasc Imaging. 2023 Apr;16(4):521-532. doi: 10.1016/j.jcmg.2022.10.023. Epub 2022 Dec 14. PMID 36648054
- [Derived] Kim HO, Jiang B, Poon EKW, Thondapu V, Kim CJ, Kurihara O, Araki M, Nakajima A, Mamon C, Dijkstra J, Lee H, Ooi A, Barlis P, Jang IK. High endothelial shear stress and stress gradient at plaque erosion persist up to 12 months. Int J Cardiol. 2022 Jun 15;357:1-7. doi: 10.1016/j.ijcard.2022.03.035. Epub 2022 Mar 16. PMID 35306029
- [Derived] Araki M, Yonetsu T, Kurihara O, Nakajima A, Lee H, Soeda T, Minami Y, Higuma T, Kimura S, Takano M, Yan BP, Adriaenssens T, Boeder NF, Nef HM, Kim CJ, McNulty I, Crea F, Kakuta T, Jang IK. Age and Phenotype of Patients With Plaque Erosion. J Am Heart Assoc. 2021 Oct 5;10(19):e020691. doi: 10.1161/JAHA.120.020691. Epub 2021 Sep 25. PMID 34569250
- [Derived] Xing L, Yamamoto E, Sugiyama T, Jia H, Ma L, Hu S, Wang C, Zhu Y, Li L, Xu M, Liu H, Bryniarski K, Hou J, Zhang S, Lee H, Yu B, Jang IK. EROSION Study (Effective Anti-Thrombotic Therapy Without Stenting: Intravascular Optical Coherence Tomography-Based Management in Plaque Erosion): A 1-Year Follow-Up Report. Circ Cardiovasc Interv. 2017 Dec;10(12):e005860. doi: 10.1161/CIRCINTERVENTIONS.117.005860. PMID 29246916